CLINICAL TRIAL: NCT00909649
Title: Influence of Fibrin Glue on Seroma Formation After Modified Radical
Brief Title: Influence of Fibrin Glue on Seroma Formation After Modified Radical Mastectomy
Acronym: MRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: mansoura university hospital, mansoura university,egypt
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: seroma in breast surgery
Record Dates: First submitted 2008-12-05; First posted 2009-05-28 (Estimated); Results first posted 2009-05-28 (Estimated); Last update posted 2009-05-28 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer
Keywords: fibrin glue; seroma; mastectomy
MeSH Terms: conditions — Breast Neoplasms; Seroma | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 fibrin glue (Active Comparator): 8 ml of fibrin glue was sprayed on the surgical area with Y canula ( doubleject application system).One milliliter of fibrin glue contains 70-100 mg. fibrinogen, 10-50 u factor 8 aprotinin 3000k iu/ml, 2-9 mg fibronectin,40-120 ug plasminogen ,4 Iu/ml thrombin, 40 mmol cocl2/L (immuno AG/austrial)
  Interventions: Procedure: fibrin glue in breast surgery
- 2 non fibrin glue (No Intervention): after good haemostasis the same sized drain was applied in axillary and breast area and incision was closed. Followed by external compression for 10 minutes in both groups. Drains were left in places until the drainage for the preceding 24 h was less than 20 ml.

INTERVENTIONS:
Procedure: fibrin glue in breast surgery — fibrin glue 8 ml in the bed after modified radical mastectomy in fibrin treated group
  Other Names: fibrin glue after modifed radical mastectomy
  Arms: 1 fibrin glue

SUMMARY:
This study was carried out from January 2005 to December 2007 at Mansoura university hospital. Fifty patients who had breast cancer were included in the study, MRM was done for all patients. Patients were randomly divided into two groups. Group І with fibrin glue 4ml of fibrin glue was sprayed on the surgical area with Y canula and group П without fibrin glue. Preoperative, Operative and Postoperative data were collected including postoperative measurement of drainage, date of removal of the drain, state of the wound, incidence of Seroma formation.

DETAILED DESCRIPTION:
This study was carried out from January 2005 to December 2007 at Mansoura university hospital, Departement 8 of surgical department. This study approved by local ethical committee Fifty patients had breast cancer were included in the study. Patients who received preoperative chemotherapy and radiotherapy were exclude Also, patients with previous axillary surgery or patients who underwent simultaneous reconstructive surgery and breast conservative surgery and locally advanced breast cancer were exclude.

Informed written consent was obtained from all patients included in the study. All patients include in the study, MRM was done for then and axillary lymphadenectomy extended to the axillary level III was done with sharp dissection and ligation of the visible lymph vessels and minor blood vessel. After performing hemostasis in the mastectomy and axillary area. .Patients were randomly divided by closed envelop into two groups. Patients were randomized at end of surgical procedure to avoid possible treatment bias during surgical procedure.

Group І (with fibrin glue) and group П without fibrin glue. In fibrin glue group. 4 ml of fibrin glue was sprayed on the surgical area with Y canula (doubleject application system). In group 11 after good haemostasis the same sized drain was applied in axillary and breast area and incision was closed. Followed by external compression for 10 minutes in both groups. Drains were left in places until the drainage for the preceding 24 h was less than 30 ml/day.

Data collected Preoperative data collected included age, body mass indexed (BMI), medical and surgical history, history of chemotherapy, radiotherapy Operative data included estimated blood loss, types of dissection, duration of the operation Postoperative data included hospital stay , postoperative measurement of drainage daily , date of removal , state of the wound ( infection , haematoma, necrosis , opened wound ), number of axillary lymph nodes dissected , cancer stage , number of axillary lymph nodes positive, incidence of Seroma formation , interval of Seroma resolution , Seroma aspirated volume and number of postoperative visits Seroma formation was defined as inability to remove participant drain by postoperative day 10 because of high output (more than 30 ml /day drain Seroma) and / or the need to aspirate of fluid after removal of the drain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with operable breast cancer

Exclusion Criteria:

* Patients who received preoperative chemotherapy and radiotherapy were exclude
* Patients with previous axillary surgery
* Patients who underwent simultaneous reconstructive surgery and breast conservative surgery
* Locally advanced breast cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ayman elnakeeb, Principal Investigator — Mansoura University Hospital
Locations (2):
- Egypt (2):
  - Ayman Elnakeeb, Mansoura , Egypt, Mansoura,egypt
  - Ayman Elnakeeb, Al Mansurah, Mansoura

REFERENCES:
- [Background] Ulusoy AN, Polat C, Alvur M, Kandemir B, Bulut F. Effect of fibrin glue on lymphatic drainage and on drain removal time after modified radical mastectomy: a prospective randomized study. Breast J. 2003 Sep-Oct;9(5):393-6. doi: 10.1046/j.1524-4741.2003.09506.x. PMID 12968960
- [Result] Johnson L, Cusick TE, Helmer SD, Osland JS. Influence of fibrin glue on seroma formation after breast surgery. Am J Surg. 2005 Mar;189(3):319-23. doi: 10.1016/j.amjsurg.2005.01.004. PMID 15792759

RESULTS

PARTICIPANT FLOW:
Recruitment Details: medical clinic
Period: Overall Study
Arm/Group | Fibrin Group | Non Fibrin Group
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibrin Group | Non Fibrin Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 22 | 22 | 44.0
  >=65 years | 3 | 3 | 6.0
Age Continuous [Mean (Standard Deviation); unit: years] | 52.2 (11.5) | 51.6 (10.8) | 51.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50.0
  Male | 0 | 0 | 0.0
Region of Enrollment [Number; unit: participants]
  Egypt | 25 | 25 | 50.0

OUTCOME MEASURES:

1. Primary Outcome: Seroma Formation
Description: the mean total drainage volume
Time Frame: within 30 days postoperative
Population: ITT
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Fibrin Group | Non Fibrin Group
Number analyzed (Participants) | 25 | 25
ml | 770.48 (70.81) | 1089.51 (75.8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No